CLINICAL TRIAL: NCT04495231
Title: Association Between Enhanced Sympathetic Activity and Cardiometabolic Complications: a Cross-sectional Study on Predictive Power of 24-hour Urinary Metanephrines (SYMPACT)
Brief Title: Sympathetic Activity and Cardiometabolic Complications
Acronym: SYMPACT
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mauro Maccario, Medical Doctor, Professor, University of Turin, Italy
Other Study IDs: SympAct 1
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Catecholamine; Overproduction; Catecholamine; Secretion; Metabolic Syndrome; Hypertensive Heart Disease; Hypertensive Kidney Disease; Diabetes Mellitus, Type 2; Hypertension,Essential
Keywords: Normetanephrine; Metanephrine; Sympathetic Nervous System; Cardiovascular System; Cardiometabolic Complications; Catecholamine; Overproduction; Catecholamine; Secretion; Metabolic Syndrome; Hypertensive Heart Disease; Hypertensive Kidney Disease; Diabetes Mellitus, Type 2; Hypertension,Essential
MeSH Terms: conditions — Metabolic Syndrome; Hypertensive Nephropathy; Diabetes Mellitus, Type 2; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent studies on catecholamine physiology have shown a direct correlation with arterial hypertension, overcoming the exclusive role in the diagnosis and follow-up of chromaffin tumors.

Nevertheless, in literature, few studies explore and reveal the utility of testing metanephrines for the evaluation of sympathetic activity and its associated cardiometabolic complications in patients with essential hypertension.

DETAILED DESCRIPTION:
Catecholamines (noradrenaline, adrenaline and dopamine) are adaptive and maladaptive stress hormones.

In the classic "fight or flight" mechanism, they activate behavioral and physiological processes that facilitate the overcoming of stress; for instance, challenged by a physical stressor, an organism responds to the threat either fighting and prevailing or accepting defeat and fleeing in avoidance.

In the pathological context, an excessive catecholamine secretion is typical of the chromaffin tissue tumors, determining a clinical picture characterized by blood pressure elevation, tachycardia, anxiety, pallor, sweating and headache.

COMT enzyme catalyzes the O-methylation of the 3-hydroxyl group of catecholamines. The O-methylated derivatives of noradrenaline, adrenaline and dopamine are normetanephrine, metanephrine and 3-methoxytyramine, respectively. The term "metanephrines" is generally used to collectively refer to the first two compounds.

Compared to catecholamines, metanephrines are characterized by longer half-life and more stable levels over time. Their superior accuracy for the diagnosis and follow-up of pheochromocytoma and paraganglioma (PPGL) has been widely proved.

Excluding patients with PPGL, however, metanephrines can be more broadly considered as reliable markers of the whole sympathetic system activity; therefore, their levels may be hypothesized to be associated to a higher rate of concurrent cardiometabolic complications and, if so, could be useful for the stratification of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Measurement of 24h urinary metanephrines at the laboratory of "City of Health and Science" hospital in Turin between 2007 and 2015
* Availability of contextual clinical patient data as collected in prospective registries of Piedmont region

Exclusion Criteria:

* Diagnosis of pheochromocytoma or paraganglioma (at the time of urinary metanephrines collection or within the following 5 years)
* Diagnosis of other forms of secondary hypertension
* Previous cardiovascular or cerebrovascular event
* Chronic heart failure
* eGFR < 50 ml/min (according to CKD-EPI)
* Liver cirrhosis
* Acute conditions and/or hospitalization in ICU (at the time of urinary metanephrines collection)
* Assumption of acetaminophen during the day before the 24-hour urine collection
* Therapy with labetalol
* Therapy with sotalol
* Therapy with alpha-methyldopa
* Therapy with MAO inhibitors
* Therapy with tricyclic antidepressants
* Therapy with buspirone
* Therapy with phenoxybenzamine
* Therapy with sulfasalazine
* Therapy with L-Dopa
* Therapy with sympathomimetic drugs or other vasopressors
* Alcohol abuse
* Cocaine abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who performed a 24h urinary metanephrines assay at the laboratory of "City of Health and Science" hospital in Turin between 2007 and 2015, with availability of full clinical data due to hospitalization at the same hospital contextually to the dosage or within ± 6 months. Exclusion criteria are specified in the appropriate section.
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Presence of left ventricular hypertrophy | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of the presence of left ventricular hypertrophy
Presence of chronic kidney disease | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of the presence of chronic kidney disease
Presence of type 2 diabetes mellitus | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of the presence of type 2 diabetes mellitus
Presence of metabolic syndrome | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of the presence of metabolic syndrome

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of systolic blood pressure values (mmHg)
Diastolic blood pressure (DBP) | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of diastolic blood pressure values (mmHg)
Resting heart rate | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of resting heart rate (bpm)
eGFR | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of eGFR values (ml/min, as estimated by CKD-EPI formula)
Urinary albumin/creatinine ratio | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of albumin/creatinine ratio values (mg/mmol)
Fasting glucose | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of fasting glucose values (mg/dl)
Total cholesterol | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of total cholesterol values (mg/dl)
HDL cholesterol | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of HDL cholesterol values (mg/dl)
LDL cholesterol | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of LDL cholesterol values (mg/dl, as estimated by Friedewald formula)
Triglycerides | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of triglycerides values (mg/dl)
Body Mass Index (BMI) | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of BMI values (kg/m2)
Cardiovascular risk as estimated by Framingham Risk Score (FRS) | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of cardiovascular risk as estimated by FRS; FRS is expressed as a percentage, with higher values indicating higher risk; patients in which the risk estimation is not applicable will be excluded from the analysis
Cardiovascular risk as estimated by Systematic COronary Risk Evaluation (SCORE) | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of cardiovascular risk as estimated by SCORE; SCORE is expressed as a percentage, with higher values indicating higher risk; patients in which the risk estimation is not applicable will be excluded from the analysis
Cardiovascular risk as estimated by Progetto Cuore Score (english translation: "Heart Project Score") | At baseline
  The value of urinary metanephrines will be evaluated as a possible predictor of cardiovascular risk as estimated by Progetto Cuore Score; Progetto Cuore Score is expressed as a percentage, with higher values indicating higher risk; patients in which the risk estimation is not applicable will be excluded from the analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maccario, MD, Principal Investigator — Endocrinology, Diabetology and Metabolism; University of Turin; Ezio Ghigo, MD, Study Chair — Endocrinology, Diabetology and Metabolism; University of Turin
Locations (1):
- Division of Endocrinology, Diabetology and Metabolism; University of Turin, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ton QV, Hammes SR. Recent insights on circulating catecholamines in hypertension. Curr Hypertens Rep. 2014 Dec;16(12):498. doi: 10.1007/s11906-014-0498-9. PMID 25304108
- [Background] Esler M. The sympathetic nervous system in hypertension: back to the future? Curr Hypertens Rep. 2015 Feb;17(2):11. doi: 10.1007/s11906-014-0519-8. PMID 25680900
- [Background] Coulson JM. The relationship between blood pressure variability and catecholamine metabolites: a pilot study. J Hum Hypertens. 2015 Jan;29(1):50-2. doi: 10.1038/jhh.2014.23. Epub 2014 Apr 3. PMID 24694800
- [Background] Lenders JW, Duh QY, Eisenhofer G, Gimenez-Roqueplo AP, Grebe SK, Murad MH, Naruse M, Pacak K, Young WF Jr; Endocrine Society. Pheochromocytoma and paraganglioma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Jun;99(6):1915-42. doi: 10.1210/jc.2014-1498. PMID 24893135
- [Background] Okuyama Y, Sakata Y. [Device treatment approaches targeting the sympathetic nervous system in patients with resistant hypertension]. Nihon Rinsho. 2015 Nov;73(11):1857-63. Japanese. PMID 26619659
- [Background] Grassi G, Mark A, Esler M. The sympathetic nervous system alterations in human hypertension. Circ Res. 2015 Mar 13;116(6):976-90. doi: 10.1161/CIRCRESAHA.116.303604. PMID 25767284
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Sever PS, Poulter NR. Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. Lancet. 2010 Mar 13;375(9718):895-905. doi: 10.1016/S0140-6736(10)60308-X. PMID 20226988
- [Background] Esler M, Lambert G, Jennings G. Increased regional sympathetic nervous activity in human hypertension: causes and consequences. J Hypertens Suppl. 1990 Dec;8(7):S53-7. PMID 1965656
- [Background] Eisenhofer G, Kopin IJ, Goldstein DS. Catecholamine metabolism: a contemporary view with implications for physiology and medicine. Pharmacol Rev. 2004 Sep;56(3):331-49. doi: 10.1124/pr.56.3.1. PMID 15317907
- [Background] Tank AW, Lee Wong D. Peripheral and central effects of circulating catecholamines. Compr Physiol. 2015 Jan;5(1):1-15. doi: 10.1002/cphy.c140007. PMID 25589262
- [Background] Goldstein DS, Eisenhofer G, Kopin IJ. Sources and significance of plasma levels of catechols and their metabolites in humans. J Pharmacol Exp Ther. 2003 Jun;305(3):800-11. doi: 10.1124/jpet.103.049270. Epub 2003 Mar 20. PMID 12649306
- [Background] Eisenhofer G, Friberg P, Pacak K, Goldstein DS, Murphy DL, Tsigos C, Quyyumi AA, Brunner HG, Lenders JW. Plasma metadrenalines: do they provide useful information about sympatho-adrenal function and catecholamine metabolism? Clin Sci (Lond). 1995 May;88(5):533-42. doi: 10.1042/cs0880533. PMID 7614812
- [Background] Masuo K, Kawaguchi H, Mikami H, Ogihara T, Tuck ML. Serum uric acid and plasma norepinephrine concentrations predict subsequent weight gain and blood pressure elevation. Hypertension. 2003 Oct;42(4):474-80. doi: 10.1161/01.HYP.0000091371.53502.D3. Epub 2003 Sep 2. PMID 12953019
- [Background] Dudenbostel T, Acelajado MC, Pisoni R, Li P, Oparil S, Calhoun DA. Refractory Hypertension: Evidence of Heightened Sympathetic Activity as a Cause of Antihypertensive Treatment Failure. Hypertension. 2015 Jul;66(1):126-33. doi: 10.1161/HYPERTENSIONAHA.115.05449. Epub 2015 May 18. PMID 25987662
- [Background] Flaa A, Aksnes TA, Kjeldsen SE, Eide I, Rostrup M. Increased sympathetic reactivity may predict insulin resistance: an 18-year follow-up study. Metabolism. 2008 Oct;57(10):1422-7. doi: 10.1016/j.metabol.2008.05.012. PMID 18803948
- [Background] Masuo K, Mikami H, Ogihara T, Tuck ML. Sympathetic nerve hyperactivity precedes hyperinsulinemia and blood pressure elevation in a young, nonobese Japanese population. Am J Hypertens. 1997 Jan;10(1):77-83. doi: 10.1016/s0895-7061(96)00303-2. PMID 9008251
- [Background] Quarti Trevano F, Dell'Oro R, Biffi A, Seravalle G, Corrao G, Mancia G, Grassi G. Sympathetic overdrive in the metabolic syndrome: meta-analysis of published studies. J Hypertens. 2020 Apr;38(4):565-572. doi: 10.1097/HJH.0000000000002288. PMID 32132429
- [Background] Mancia G, Bousquet P, Elghozi JL, Esler M, Grassi G, Julius S, Reid J, Van Zwieten PA. The sympathetic nervous system and the metabolic syndrome. J Hypertens. 2007 May;25(5):909-20. doi: 10.1097/HJH.0b013e328048d004. PMID 17414649
- [Background] Straznicky NE, Grima MT, Sari CI, Karapanagiotidis S, Wong C, Eikelis N, Richards KL, Lee G, Nestel PJ, Dixon JB, Lambert GW, Schlaich MP, Lambert EA. The relation of glucose metabolism to left ventricular mass and function and sympathetic nervous system activity in obese subjects with metabolic syndrome. J Clin Endocrinol Metab. 2013 Feb;98(2):E227-37. doi: 10.1210/jc.2012-3277. Epub 2012 Dec 27. PMID 23271752
- [Background] Schlaich MP, Kaye DM, Lambert E, Sommerville M, Socratous F, Esler MD. Relation between cardiac sympathetic activity and hypertensive left ventricular hypertrophy. Circulation. 2003 Aug 5;108(5):560-5. doi: 10.1161/01.CIR.0000081775.72651.B6. Epub 2003 Jul 7. PMID 12847071
- [Background] Wang W, Mu L, Su T, Ye L, Jiang Y, Jiang L, Zhou W. Plasma Metanephrines Are Associated With Glucose Metabolism in Patients With Essential Hypertension. Medicine (Baltimore). 2015 Sep;94(37):e1496. doi: 10.1097/MD.0000000000001496. PMID 26376391
- [Background] Brown MJ, Causon RC, Barnes VF, Brennan P, Barnes G, Greenberg G. Urinary catecholamines in essential hypertension: results of 24-hour urine catecholamine analyses from patients in the Medical Research Council trial for mild hypertension and from matched controls. Q J Med. 1985 Oct;57(222):637-51. PMID 4080953
- [Background] Zhou Y, Yuan J, Wang Y, Qiao S. Plasma metanephrins are associated with myocardial hypertrophy and cardiac diastolic function in patients with essential hypertension. Clin Invest Med. 2020 Apr 5;43(1):E22-E29. doi: 10.25011/cim.v43i1.33581. PMID 32247299